CLINICAL TRIAL: NCT03246360
Title: Pharmacological Comparison of Continuous and Intermittent Infusions of Cloxacillin During Bone and Joint Infections: a Prospective, Randomized, Open-label, Monocentric Crossover Study.
Brief Title: Pharmacological Comparison of Continuous and Intermittent Infusions of Cloxacillin
Acronym: CLOXA Continue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16-PP-04
Record Dates: First submitted 2017-07-28; First posted 2017-08-11 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Infection; Methicillin Susceptible Staphylococcus Aureus Infection; Cloxacillin Treatment
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent administration of cloxacillin (Active Comparator)
  Interventions: Drug: Modification for administration mode of cloxacillin antibiotic
- continuous administration of cloxacillin (Experimental)
  Interventions: Drug: Modification for administration mode of cloxacillin antibiotic

INTERVENTIONS:
Drug: Modification for administration mode of cloxacillin antibiotic — For intermittent administration, patients will benefit from cloxacillin treatment in conventional hospitalization, in accordance with national guidelines, at a dose of 150 mg / kg per day in 4 infusions, not exceeding the maximum daily dose of 12 g / day according to.
  For continuous administration the same quantity of cloxacillin 150 mg / kg per day, without exceeding the maximum daily dose of 12 g / day, will be delivered by a self-propelled syringe in twice 12 hours. Patients randomly assigned to receive continuous administration will receive a dose of cloxacillin equivalent to the dose administered 4 times daily during iterative administration using a self-pulsating syringe. For the first day of the study, this loading dose will be subtracted from the 150 mg / kg dose to be administered continuously over the remaining 23 hours of the first day of the study and never exceed 12g / day.
  Pharmacological dosages will be performed on the third and sixth day in both arms

SUMMARY:
Our objective is to establish pharmacological equivalence of intermittent and continuous infusion of cloxacillin during methicillin-susceptible Staphylococcus aureus (MSSA) bone and joint infections (BJI). Twelve patients suffering MSSA BJI will receive both administration modalities and serum concentrations of cloxacillin will be determined after 3 days of II and 3 days of continuous infusion in a prospective, randomized, open-label, monocentric crossover study design.

DETAILED DESCRIPTION:
Introduction Staphylococcus aureus is the main causative agent of bone and joint infections (BJI). More than 80% of the strains isolated in France are methicillin-susceptible (MSSA). During the early phase of MSSA BJI management national and international guidelines recommend the use of intra-venous type M penicillin with a dosage ranging from 100 to 200 mg/kg/day. Pharmacological properties of this class of penicillin require 4 to 6 infusions by day. Continuous infusion of beta-lactams is increasingly used especially in intensive care units. It allows an improvement of pharmacokinetic/pharmacodynamics (PK/PD) parameters and a reduction in time dedicated to infusion preparations by the nurses. However pharmacological data regarding such administration is required for type M penicillin.

Design A 6-day, prospective, randomized, open-label, monocentric crossover study

Participants Twelve adult patients with MSSA BJI

Intervention Patients will be randomized in two groups: the first group will receive 3 days of cloxacillin (150 mg/kg/day) through 4 intermittent infusions/day followed by 3 days of cloxacillin (150 mg/kg/day) through continuous infusion (2 infusions during 12 hours). In the second group the infusion modalities will be inverted and continuous infusion will be preceded by a loading dose. Serum concentrations of cloxacillin will be determined at Day 3 and Days 6 The area under the curve / minimal inhibitory concentration ratio will be use to establish the equivalence between both administration modalities.

ELIGIBILITY:
Inclusion Criteria:

* Staphylococcus aureus sensitive to methicillin and to be treated with cloxacillin by injectable antibiotic monotherapy For patients with Osteo-articular infection on material

  * Presence of a fistula in contact with the prosthesis or implant.
  * Pus in the joint or in contact with the prosthesis or implant
  * Presence of at least 1 positive sample (1 sampling by articular puncture or 1 peroperative sampling or by blood culture)
  * A histological analysis of the peri-prosthetic osteo-articular tissue which is the object of acute inflammation is a strong argument in favor of an Osteo-articular infection on material

For spondylodiscitis

* Culture of a disco-vertebral biopsy puncture to isolate a methicillin sensitive S. aureus
* Positive haemocultures for S. aureus sensitive to methicillin with imaging examination (CT or MRI of the spine) showing images of spondylodiscitis

For primitive arthritis :

* Culture of a positive methicillin-sensitive S. aureus articular fluid puncture
* Cultivation of a methicillin-sensitive S. aureus-positive surgical joint lavage fluid

For osteitis the diagnosis is based on the following criterion:

*Culture of surgical specimens from a focal zone of methicillin-sensitive S. aureus-positive osteitis

Exclusion Criteria:

* Allergy to betalactamines
* Taking penicillin M within 36 hours before inclusion Renal function impaired with a glomerular filtration rate measured by MDRD formula of less than 30 ml / min
* Patient with renal function expected to change within 6 days of inclusion
* Hepatocellular insufficiency, whatever the degree

  -*Methotrexate intake
* Polytransfused (more than 2 CGR) in the previous week
* Patients requiring resuscitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
The equivalence of the Pharmacokinetic-Pharmacodynamic indicators commonly used for the study of betalactamines: T> minimal inhibitory concentration | Six days
The equivalence of the Pharmacokinetic-Pharmacodynamic indicators commonly used for the study of betalactamines: the area under the curve (AUC) / minimal inhibitory concentration | Six days

CONTACTS AND LOCATIONS:
Overall Officials: Johan Johan, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No